CLINICAL TRIAL: NCT00027326
Title: Collection of Peripheral Blood and/or Urine From Patients Undergoing Radiation Therapy
Brief Title: Collection of Blood and Urine From Patients Undergoing Radiation Therapy
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020064; 02-C-0064; NCT00995943 (obsolete NCT alias)
Record Dates: First submitted 2006-07-13; First posted 2001-12-03 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12-16

CONDITIONS: Carcinoma; Cancer; Tumor
Keywords: Blood; Samples; Radiation; Urine; Cancer; Natural History
MeSH Terms: conditions — Carcinoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Patients: Candidate for or currently receiving radiotherapy

SUMMARY:
Background:

-Research in NCI's Radiation Oncology Branch depends on the availability of blood and urine samples from patients receiving radiation therapy.

Objectives:

-To explore the effects of radiation therapy on gene expression in white blood cells, to measure radiation damage in red blood cells and to examine changes in hormone levels in the blood and urine after radiation therapy.

Eligibility:

-Patients 18 years of age and older who are receiving radiation therapy.

Design:

* Blood and urine samples are collected when participants enter the study.
* Additional samples may be collected at different times during and after treatment. Ideally, samples are obtained before, at the completion of, and 1 month following radiation therapy. Blood samples usually will be collected during routine patient monitoring procedures and will not require an additional needle stick.
* A total of 300 patients will be studied at the NCI in Bethesda, MD, Johns Hopkins University in Baltimore and the University of Pennsylvania in Philadelphia.

DETAILED DESCRIPTION:
BACKGROUND:

Evolving research initiatives in the Radiation Oncology Branch (ROB) NCI, depend upon the availability of blood and urine samples from patients receiving radiotherapy.

Examples of planned studies include an exploration of the effects of radiotherapy on peripheral leukocyte phenotype, peripheral blood protein and metabolism changes as well as measurements of matrix metalloproteinases (MMP) in urine.

OBJECTIVES:

This protocol provides a means of acquiring blood and urine samples in patients receiving radiation therapy for a variety of conditions.

ELIGIBILITY:

Patients seen in the radiation oncology clinic will be asked to donate blood and/or urine before, during and after their treatment.

DESIGN:

This is a pilot, exploratory study to evaluate the effects of ionizing radiation in blood and/ or urine.

On most occasions, the blood samples will be obtained as a component of routine patient monitoring and will not necessitate an additional venipuncture.

Blood and urine samples will be processed and stored in the Radiation Oncology Branch and Basic Research Laboratory, CCR, NCI, for use in the research efforts of the branch.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must be co-enrolled in a NIH CC protocol in which radiation will be administered.
  2. Patients must be a candidate for, or currently receiving radiotherapy.
  3. Age greater than or equal to 18 years.
  4. Ability of subject or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Patients who have unobtainable data regarding previous radiation therapy.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients currently a candidate or currently receiving radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2001-12-02 (Actual)

PRIMARY OUTCOMES:
To acquire peripheral blood and/or urine samples from patients receiving radiation therapy in the Radiation Oncology Branch, NCI. | At the time of the enrollment, a blood and/or a urine sample will be collected. Blood and/or urine will also be collected at the completion of radiotherapy and at 1 month follow- up.
  collection of blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-C-0064.html